CLINICAL TRIAL: NCT03784872
Title: Laparoscopic Ventrosuspension for Women With Retroverted Uterus and Pelvic Pain Syndromes: A New Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic guided Ventrosuspension — Laparoscopy was done. Under vision the skin overlying the attachment of the round ligament to the anterior abdominal wall was incised followed by introduction of 30 curved needle attached to absorpable Vicryl 2/0 suture through the incision and withdrawn through grasper under laparoscopi vision. The needle was turned around the round ligament all through its length to plicate it then the needle was pushed again beside its entry side to appear at the skin incision. The same was repeated on the other side and both sutures were tied at the subcutaneous tissue simultaneously. then the laparoscopy was withdrawn followed by closure of the skin incision.

SUMMARY:
In women with retroverted retroverted uterus complaining of pelvic pain, Laparoscopy was done. Under vision the skin overlying the attachment of the round ligament to the anterior abdominal wall was incised followed by introduction of 30 curved needle attached to absorpable Vicryl 2/0 suture through the incision and withdrawn through grasper under laparoscopi vision. The needle was turned around the round ligament all through its length to plicate it then the needle was pushed again beside its entry side to appear at the skin incision. The same was repeated on the other side and both sutures were tied at the subcutaneous tissue simultaneously. then the laparoscopy was withdrawn followed by closure of the skin incision.

DETAILED DESCRIPTION:
In women with retroverted retroverted uterus complaining of pelvic pain, Laparoscopy was done. Under vision the skin overlying the attachment of the round ligament to the anterior abdominal wall was incised followed by introduction of 30 curved needle attached to absorpable Vicryl 2/0 suture through the incision and withdrawn through grasper under laparoscopi vision. The needle was turned around the round ligament all through its length to plicate it then the needle was pushed again beside its entry side to appear at the skin incision. The same was repeated on the other side and both sutures were tied at the subcutaneous tissue simultaneously. then the laparoscopy was withdrawn followed by closure of the skin incision using Vicryl 2/0 suture.

ELIGIBILITY:
Inclusion Criteria:

* women with chronic pelvic pain for more than 6 months duration
* women with retroverted retroflexed uterus
* no response to analgesics
* fit for laparoscopic surgery

Exclusion Criteria:

* Women with other causes of pelvic pain as ovarian cysts
* women with neurological disorders
* psychologically disturbed,
* Women with systemic or pelvic infections,

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: VAS | 6 months after the operation
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided